CLINICAL TRIAL: NCT05311774
Title: Efficacy of Duloxetine in Conjunction With Tramadol for Chronic Cancer Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Madona M.NOMAN, Doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Duloxetine in cancer pain
Record Dates: First submitted 2022-03-15; First posted 2022-04-05 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Cancer Pain
Keywords: duloxetine; tramadol; cancer pain
MeSH Terms: conditions — Cancer Pain | interventions — Duloxetine Hydrochloride; Tramadol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- •tramadol and duloxetine (Experimental): patients will receive tramadol 50 mg twice daily, titration will be done every 3days until 2 weeks, maximum dose will be 400mg daily and will receive duloxetine 30mg daily fixed dose in combination with tramadol. Investigators will follow up the patients for 3 months
  Interventions: Drug: Duloxetine 30 mg; Drug: Tramadol
- tramadol and placebo (Active Comparator): patients will receive tramadol 50 mg twice daily, titration will be done every 3days until 2 weeks, maximum dose will be 400mg daily and will receive placebo drug once daily in combination with tramadol. Investigators will follow up the patients for 3 months
  Interventions: Drug: Tramadol; Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine 30 mg — tablet
  Other Names: cymbatex 30 mg
  Arms: •tramadol and duloxetine
Drug: Tramadol — tablet
  Other Names: amadol
Drug: Placebo — tablet
  Arms: tramadol and placebo

SUMMARY:
Cancer pain is one of the most common and problematic symptoms. Opioids are typically the most common drugs used in the treatment of cancer pain,they are limited due to their side effects.

Tramadol is a centrally acting non-opiate analgesic with low affinity for μ-opioid receptors, and is effective in the treatment of moderate to severe pain.

Neuropathic pain is typically not amenable to standard opiate therapy, and the addition of tricyclic antidepressants or/and antiepileptic drugs can offer a very effective treatment strategy in such patients.

Duloxetine is a Serotonin Norepinephrine Reuptake Inhibitor (SNRI) that has been used traditionally for its antidepressant qualities and has also analgesic benefit in the treatment of neuropathic pain. Duloxetine exerts its analgesic action through central and peripheral pain modulation .

DETAILED DESCRIPTION:
Cancer pain is one of the most common and problematic symptoms.uncontrolled pain affect quality of life and daily activities .Cancer pain has two main categories nociceptive and neuropathic pain,Cancer pain is often a combination of nociceptive and neuropathic pain.

A framework for managing pain often starts with the World Health Organization (WHO) Analgesic Ladder, step 1 use non opioid analgesics, step 2 weak opioids, step 3 strong opioids, step 4 interventions non pharmacological, adjuvants can be added to any step .

Opioids are typically the most common drugs used in the treatment of cancer pain. They work by binding to μ-opioid receptors within the central nervous system, which are responsible for opioid mediated analgesia, respiratory depression, sedation, physiological dependence, and tolerance, they are limited due to their side effects as nausea, constipation, sedation, and confusion, prolonged use of opioids may lead to development of tolerance, abnormal hypersensitivity to pain.

Tramadol is a centrally acting non-opiate analgesic with low affinity for μ-opioid receptors, and is effective in the treatment of moderate to severe pain. It has been also shown to inhibit reuptake of serotonin and norepinephrine, which synergistically enhances its weak opioid mechanism of action.

This may explain the reduced incidences of abuse, respiratory depression and other adverse effects of traditional opioids in patients on long-term tramadol therapy.it is a useful drug in patients with cancer pain both with nociceptive and neuropathic pain .Neuropathic pain is typically not amenable to standard opiate therapy, and the addition of tricyclic antidepressants or/and antiepileptic drugs can offer a very effective treatment strategy in such patients.

Adjuvant analgesics are drugs primarily marketed for other indications, such as depression, but also have an important role in cancer pain management. Antidepressants, such as serotonin- norepinephrine reuptake inhibitors (duloxetine, venlafaxine) or tricyclics ( nortriptyline, amitriptyline) and anticonvulsants (pregabalin, gabapentin, carbamazepine) have efficacy in the treatment of pain, particularly neuropathic pain .Duloxetine is a Serotonin Norepinephrine Reuptake Inhibitor (SNRI) that has been used traditionally for its antidepressant qualities and has also analgesic benefit in the treatment of neuropathic pain . Duloxetine exerts its analgesic action through central and peripheral pain modulation , it enhances the effect of serotonin and norepinephrine on descending inhibitory pain pathways in the brain and spinal cord and activation of some cerebral prefrontal areas . Besides, it has been claimed that Duloxetine has an anti-nociceptive effect through Na + channel block , therefore it suppresses the neuronal cell firing resulting from peripheral injury . The most common adverse effects of duloxetine, which may lead to discontinuation of the drug, are nausea, dizziness, and somnolence .There is a possibility that duloxetine was effective in both activation of the descending pain modulatory system and the improvement of depressive mood, the effect may have partly taken place due to elevation of the pain threshold through the antidepressant effect of duloxetine . Recently, the efficacy of duloxetine has been reported in patients with chemotherapy-induced peripheral neuropathy (CIPN) and in non-cancer neuropathic pain. .

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer pain

  1. age from 20-70 years old.
  2. not receiving any type of analgesia before (opioid naïve, no adjuvants).

Exclusion Criteria:

1. Difficult to be assessed for pain.
2. Any contraindication for duloxetine or tramadol.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
concentration of tramadol consumption | at one month
  all participants(400 patients) will receive tramadol 50 mg twice daily, titration will be done every 3days until 2 weeks,according to changes in visual analogue scale for pain maximum dose will be 400mg daily, one group of participants(200 patients) will receive duloxetine 30mg daily fixed dose in combination with tramadol,decrease in concentration of tramadol consumption means better results,the other group(200 patients) will receive placebo drug once daily in combination with tramadol.

SECONDARY OUTCOMES:
concentration of tramadol consumption | at 2 month and 3 month
  all participants(400 patients) will receive tramadol 50 mg twice daily, titration will be done according to changes in visual analogue scale for pain, maximum dose will be 400mg daily, one group of participants(200 patients) will receive duloxetine 30mg daily fixed dose in combination with tramadol,decrease in concentration of tramadol consumption means better results,the other group(200 patients) will receive placebo drug once daily in combination with tramadol.
- change in pain with visual analogue scale | at 3,6,9 and 12 days , 2 weeks,1 month,2 month,3 month
  subjective scale by the participants for pain intensity from 0 to 10, minimum value is zero that means no pain, maximum value is 10 that means unbearable pain, higher scores mean worse outcome
type of pain that relieved better | at 1 month,2 month and 3 month
  type of pain that responds better to duloxetine and tramadol (neuropathic or nociceptive), using visual analogue scale for pain intensity (subjective scale by the participants for pain intensity from 0 to 10, minimum value is zero that means no pain, maximum value is 10 that means unbearable pain, higher scores mean worse outcome)
Leeds Assessment of Neuropathic Symptoms and Signs Scale if neuropathic pain | at 1 month,2 month and 3 month
  used for neuropathic pain consists of seven questions minimum value 0 ,maximum value 24,scoring a score of 12 or more suggests pain of predominantly neuropathic origin
Scale Assessing Pain Intensity and Interference (Pain, Enjoyment, General Activity) | at 1 month,2 month and 3 month
  consisting of three questions for the participant,responses from 0 to 10 ,responses to three questions added then divided by three to get a mean score out of ten
Depression scores by the Patient Health Questionnaire | at 1 month,2 month and 3 month
  consists of 9 questions for the participant ,This is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of "not at all," "several days," "more than half the days," and "nearly every day," respectively, total score for the nine items ranges from 0 to 27,higher scores means worse outcome
Anxiety scores by the Patient Health Questionnaire | at 1 month,2 month and 3 month
  consists of 7 questions for the participant ,This is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of "not at all," "several days," "more than half the days," and "nearly every day," respectively, total score for the seven items ranges from 0 to 21,higher scores means worse outcome
Flanagan Quality of Life Scale | at 1 month,2 month and 3 month
  consists of 16 items ,seven responses are delighted(7),pleased(6),mostly satisfied(5),mixed(4),mostly dissatisfied (3),unhappy(2),terrible(1),ranging from 16 to 112,average for healthy 90
Side effects as nausea, vomiting, constipation, sedation, arrhythmia and hypertension | up to 3 month
  participants will be asked about side effects from duloxetine as nausea,vomiting, constipation, sedation, (onset,duration,offset, bearable or not ,affecting quality of life), arrhythmia (type of arrhythmia from electrocardiogram ,onset,duration,offset),hypertension (by measuring blood pressure ,onset ,duration ,offset)

CONTACTS AND LOCATIONS:
Overall Officials: khaled M Fares, MD, Study Director — Assiut University; Ahmad M Abd EL Rahman, MD, Study Director — Assiut University; Diab F Hetta, MD, Study Director — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van den Beuken-van Everdingen MH, Hochstenbach LM, Joosten EA, Tjan-Heijnen VC, Janssen DJ. Update on Prevalence of Pain in Patients With Cancer: Systematic Review and Meta-Analysis. J Pain Symptom Manage. 2016 Jun;51(6):1070-1090.e9. doi: 10.1016/j.jpainsymman.2015.12.340. Epub 2016 Apr 23. PMID 27112310
- [Background] Greco MT, Roberto A, Corli O, Deandrea S, Bandieri E, Cavuto S, Apolone G. Quality of cancer pain management: an update of a systematic review of undertreatment of patients with cancer. J Clin Oncol. 2014 Dec 20;32(36):4149-54. doi: 10.1200/JCO.2014.56.0383. Epub 2014 Nov 17. PMID 25403222
- [Background] Ashby MA, Fleming BG, Brooksbank M, Rounsefell B, Runciman WB, Jackson K, Muirden N, Smith M. Description of a mechanistic approach to pain management in advanced cancer. Preliminary report. Pain. 1992 Nov;51(2):153-161. doi: 10.1016/0304-3959(92)90256-B. PMID 1283009
- [Background] Knudsen AK, Aass N, Fainsinger R, Caraceni A, Klepstad P, Jordhoy M, Hjermstad MJ, Kaasa S. Classification of pain in cancer patients--a systematic literature review. Palliat Med. 2009 Jun;23(4):295-308. doi: 10.1177/0269216309103125. Epub 2009 Mar 13. PMID 19286741
- [Background] . World Health Organization. Cancer Pain Relief. 2. Geneva: WHO; 1996. 7.
- [Background] Gutstein HB, Akil H. Opioid analgesics. In: Hardman JG, Limbrid E, editors. Goodman and Gilman's the Pharmacological Basis of Therapeutics. 10. New York: McGraw-Hill Professional; 2001. pp. 569-619.
- [Background] Alvarez V, Arttamangkul S, Williams JT. A RAVE about opioid withdrawal. Neuron. 2001 Dec 6;32(5):761-3. doi: 10.1016/s0896-6273(01)00530-x. PMID 11738021
- [Background] Raffa RB, Friderichs E, Reimann W, Shank RP, Codd EE, Vaught JL. Opioid and nonopioid components independently contribute to the mechanism of action of tramadol, an 'atypical' opioid analgesic. J Pharmacol Exp Ther. 1992 Jan;260(1):275-85. PMID 1309873
- [Background] Desmeules JA, Piguet V, Collart L, Dayer P. Contribution of monoaminergic modulation to the analgesic effect of tramadol. Br J Clin Pharmacol. 1996 Jan;41(1):7-12. doi: 10.1111/j.1365-2125.1996.tb00152.x. PMID 8824687
- [Background] Raffa RB. Pharmacology of oral combination analgesics: rational therapy for pain. J Clin Pharm Ther. 2001 Aug;26(4):257-64. doi: 10.1046/j.1365-2710.2001.00355.x. PMID 11493367
- [Background] Russell IJ, Kamin M, Bennett RM, Schnitzer TJ, Green JA, Katz WA. Efficacy of tramadol in treatment of pain in fibromyalgia. J Clin Rheumatol. 2000 Oct;6(5):250-7. doi: 10.1097/00124743-200010000-00004. PMID 19078481
- [Background] Arbaiza D, Vidal O. Tramadol in the treatment of neuropathic cancer pain: a double-blind, placebo-controlled study. Clin Drug Investig. 2007;27(1):75-83. doi: 10.2165/00044011-200727010-00007. PMID 17177582
- [Background] Duhmke RM, Cornblath DD, Hollingshead JR. Tramadol for neuropathic pain. Cochrane Database Syst Rev. 2004;(2):CD003726. doi: 10.1002/14651858.CD003726.pub2. PMID 15106216
- [Background] Finnerup NB, Attal N, Haroutounian S, McNicol E, Baron R, Dworkin RH, Gilron I, Haanpaa M, Hansson P, Jensen TS, Kamerman PR, Lund K, Moore A, Raja SN, Rice AS, Rowbotham M, Sena E, Siddall P, Smith BH, Wallace M. Pharmacotherapy for neuropathic pain in adults: a systematic review and meta-analysis. Lancet Neurol. 2015 Feb;14(2):162-73. doi: 10.1016/S1474-4422(14)70251-0. Epub 2015 Jan 7. PMID 25575710
- [Background] Collins SL, Moore RA, McQuayHJ, Wiffen P. Antidepressants and anticonvulsants for diabetic neuropathy and postherpetic neuralgia: a quantitative systematic review. J Pain Symptom Manage. 2000 Dec;20(6):449-58. doi: 10.1016/s0885-3924(00)00218-9. PMID 11131263
- [Background] McMenamin E. Pain management principles. Curr Probl Cancer. 2011 Nov-Dec;35(6):317-24. doi: 10.1016/j.currproblcancer.2011.10.006. No abstract available. PMID 22136705
- [Background] Verdu B, Decosterd I, Buclin T, Stiefel F, Berney A. Antidepressants for the treatment of chronic pain. Drugs. 2008;68(18):2611-32. doi: 10.2165/0003495-200868180-00007. PMID 19093703
- [Background] Dworkin RH, O'Connor AB, Backonja M, Farrar JT, Finnerup NB, Jensen TS, Kalso EA, Loeser JD, Miaskowski C, Nurmikko TJ, Portenoy RK, Rice ASC, Stacey BR, Treede RD, Turk DC, Wallace MS. Pharmacologic management of neuropathic pain: evidence-based recommendations. Pain. 2007 Dec 5;132(3):237-251. doi: 10.1016/j.pain.2007.08.033. Epub 2007 Oct 24. PMID 17920770
- [Background] Quilici S, Chancellor J, Lothgren M, Simon D, Said G, Le TK, Garcia-Cebrian A, Monz B. Meta-analysis of duloxetine vs. pregabalin and gabapentin in the treatment of diabetic peripheral neuropathic pain. BMC Neurol. 2009 Feb 10;9:6. doi: 10.1186/1471-2377-9-6. PMID 19208243
- [Background] Onutu AH. Duloxetine, an antidepressant with analgesic properties - a preliminary analysis. Rom J Anaesth Intensive Care. 2015 Oct;22(2):123-128. PMID 28913467
- [Background] Basbaum AI, Fields HL. Endogenous pain control systems: brainstem spinal pathways and endorphin circuitry. Annu Rev Neurosci. 1984;7:309-38. doi: 10.1146/annurev.ne.07.030184.001521. No abstract available. PMID 6143527
- [Background] Jones CK, Peters SC, Shannon HE. Efficacy of duloxetine, a potent and balanced serotonergic and noradrenergic reuptake inhibitor, in inflammatory and acute pain models in rodents. J Pharmacol Exp Ther. 2005 Feb;312(2):726-32. doi: 10.1124/jpet.104.075960. Epub 2004 Oct 19. PMID 15494550
- [Background] Wang SY, Calderon J, Kuo Wang G. Block of neuronal Na+ channels by antidepressant duloxetine in a state-dependent manner. Anesthesiology. 2010 Sep;113(3):655-65. doi: 10.1097/ALN.0b013e3181e89a93. PMID 20693878
- [Background] Nakajima K, Obata H, Iriuchijima N, Saito S. An increase in spinal cord noradrenaline is a major contributor to the antihyperalgesic effect of antidepressants after peripheral nerve injury in the rat. Pain. 2012 May;153(5):990-997. doi: 10.1016/j.pain.2012.01.029. Epub 2012 Mar 15. PMID 22424692
- [Background] Allgulander C, Nutt D, Detke M, Erickson J, Spann M, Walker D, Ball S, Russell J. A non-inferiority comparison of duloxetine and venlafaxine in the treatment of adult patients with generalized anxiety disorder. J Psychopharmacol. 2008 Jun;22(4):417-25. doi: 10.1177/0269881108091588. PMID 18635722
- [Background] Colleoni M, Mandala M, Peruzzotti G, Robertson C, Bredart A, Goldhirsch A. Depression and degree of acceptance of adjuvant cytotoxic drugs. Lancet. 2000 Oct 14;356(9238):1326-7. doi: 10.1016/S0140-6736(00)02821-X. PMID 11073026
- [Background] McDonald MV, Passik SD, Dugan W, Rosenfeld B, Theobald DE, Edgerton S. Nurses' recognition of depression in their patients with cancer. Oncol Nurs Forum. 1999 Apr;26(3):593-9. PMID 10214600
- [Background] Meyer HA, Sinnott C, Seed PT. Depressive symptoms in advanced cancer. Part 2. Depression over time; the role of the palliative care professional. Palliat Med. 2003 Oct;17(7):604-7. doi: 10.1191/0269216303pm813oa. PMID 14594151
- [Background] Bouhassira D, Wilhelm S, Schacht A, Perrot S, Kosek E, Cruccu G, Freynhagen R, Tesfaye S, Lledo A, Choy E, Marchettini P, Mico JA, Spaeth M, Skljarevski V, Tolle T. Neuropathic pain phenotyping as a predictor of treatment response in painful diabetic neuropathy: data from the randomized, double-blind, COMBO-DN study. Pain. 2014 Oct;155(10):2171-9. doi: 10.1016/j.pain.2014.08.020. Epub 2014 Aug 27. PMID 25168665
- [Background] Smith EM, Pang H, Cirrincione C, Fleishman S, Paskett ED, Ahles T, Bressler LR, Fadul CE, Knox C, Le-Lindqwister N, Gilman PB, Shapiro CL; Alliance for Clinical Trials in Oncology. Effect of duloxetine on pain, function, and quality of life among patients with chemotherapy-induced painful peripheral neuropathy: a randomized clinical trial. JAMA. 2013 Apr 3;309(13):1359-67. doi: 10.1001/jama.2013.2813. PMID 23549581